CLINICAL TRIAL: NCT02752399
Title: Applicability of the Six Minutes Walk Test and Shuttle Walk Test and Evaluation of Peripheral and Respiratory Muscle Function, Autonomic Control, Quality of Life and Sleep, Inflammatory Markers and Tissue Perfusion in Eisenmenger Syndrome
Brief Title: Six Minutes Walk Test and Shuttle Walk Test in Eisenmenger Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Bruna Caroline Matos Garcia, Physiotherapist, Federal University of São Paulo
Other Study IDs: 1.462.879
Record Dates: First submitted 2016-04-18; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Eisenmenger Complex; Pulmonary Hypertension; Congenital Heart Defects
MeSH Terms: conditions — Eisenmenger Complex; Hypertension, Pulmonary; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to verify the applicability Six minutes walk test and Shuttle walk test in assessing functional capacity in patients with Eisenmenger Syndrome. Patients will undergo three functional tests, being the six-minute walk test, shuttle walk test and cardiopulmonary exercise test on a cycle ergometer, associated with evaluation of metabolic and ventilatory variables and cardiac monitoring throughout the test.

DETAILED DESCRIPTION:
It has seen an increasing number of individuals with congenital heart diseases mainly due to the development of new diagnostic techniques, assessment and treatment, thereby contributing to longer survival. These individuals that survive to adulthood, many sometimes develop other secondary problems to the underlying pathology, one of Pulmonary Arterial Hypertension. The Syndrome Eisenmenger is the most advanced form of pulmonary hypertension secondary to congenital heart defects. It is known that patients with pulmonary hypertension secondary congenital heart disease have marked functional limitation and high risk of death. Among the various forms of assess exercise capacity, Walk Test Six Minutes (6MWT), Shuttle walking test and Cardiopulmonary Exercise Test are among the most applicable. Little has been studied about the patients with pulmonary hypertension secondary to congenital heart disease and Eisenmenger Syndrome. The characterization of this profile of patients against the effort becomes necessary and useful in determining strategies and identification of factors that may be limited to functional capacity and quality of life. Objectives: To verify the applicability Six minutes walk test and Shuttle walk test in assessing functional capacity in patients with Eisenmenger Syndrome. Methods: Cross-sectional study with patients diagnosed with Eisenmenger Syndrome, of both sexes, without changing pace or lower limbs, who have performed echocardiography in the last 6 months and clinical stability. Patients will undergo three functional tests, being the six-minute walk test, shuttle walk test and cardiopulmonary exercise test on a cycle ergometer, associated with evaluation of metabolic and ventilatory variables and cardiac monitoring throughout the test. Also will be held assess respiratory endurance and strength, peripheral muscle strength and manual pinch, Heart rate variability, inflammatory mediators and blood lactate, besides questionnaires about quality of life, quality of sleep and daytime drowsiness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Eisenmenger syndrome
* To understand the realization of tests
* That do ambulatory monitoring of congenital heart of Federal University of São Paulo..

Exclusion Criteria:

* Donw Syndrome
* Changing pace or lower limbs
* Neuromuscular disease
* Pulmonary Obstructive disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with eisenmenger syndrome that do ambulatory monitoring of congenital heart of Federal University of São Paulo.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Six minute walk test to measure functional capacity in eisenmenger syndrome | One day
  Six minute walk test will be done with metabolic and ventilatory monitoring and Compared to the cardiopulmonary exercise testing variables , seeing your similarity and if this first test is applicable to measurement functional capacity in Eisenmenger syndrome
Shuttle walk test to measure functional capacity in Eisenmenger syndrome | One day
  Shuttle walk test will be done with metabolic and ventilatory monitoring and Compared to the cardiopulmonary exercise testing variables , seeing your similarity and if this first test is applicable to measurement functional capacity in Eisenmenger syndrome

SECONDARY OUTCOMES:
Oxygen uptake kinetics during six minute walk test in Eisenmenger syndrome | one day
  Six minute walk test will be done with metabolic and ventilatory monitoring and we will go evaluate behavior of oxygen uptake kinetics in Eisenmenger Syndrome
Correlation between Functional capacity evaluate with six minute walk test and respiratory function evaluate with manovacuometry, spirometry and muscular respiratory endurance. | one day
Correlation between Functional capacity evaluate with six minute walk test and peripheric muscular function, evaluate with quadriceps dynamometry and strength of handgrip | one day
Correlation between Functional capacity evaluate with six minute walk test and autonomic function, evaluate with cardiofrequency | one day
Correlation between Functional capacity evaluate with six minute walk test and life quality evaluate with SF-36 health survey questionnaire | one day
Correlation between Functional capacity evaluate with six minute walk test and sleep quality, evaluate with pittsburgh questionnaire for sleep and Epworth Sleepiness Scale | one day
Correlation between Functional capacity evaluate with six minute walk test and blood inflammatory mediators and blood lactate | one day

CONTACTS AND LOCATIONS:
Overall Officials: Solange Guizilini, mastermind, Study Chair — Federal University of São Paulo
Locations (1):
- Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No